CLINICAL TRIAL: NCT05082935
Title: Optimizing SARS-CoV-2 Testing and Promotores Interventions to Serve Latinx Communities
Brief Title: COVID-19: Healthy Oregon (Oregon Saludable): Together We Can (Juntos Podemos) Phase II
Acronym: OSJP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oregon (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Leslie Leve,, Professor and Lorry Lokey Chair, College of Education; Associate Director, Prevention Science Institute; Associate Vice President for Research, University of Oregon
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 10032020.002.2; 3P50DA048756-03S3 (NIH)
Record Dates: First submitted 2021-10-15; First posted 2021-10-19 (Actual); Results first posted 2024-07-22 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: Health Behavior; Health Care Utilization
Keywords: Latinx; SARS-CoV-2; COVID-19; Hispanic; Testing; Vaccination
MeSH Terms: conditions — Health Behavior; Patient Acceptance of Health Care; COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Partner-optimized venue placement strategy (Experimental): The Phase II intervention involves outreach from community partners to attend testing at existing events organized by community partners, such as the Mexican Consulate. At the event, it includes the on-site Promotores de Salud psychoeducation related to SARS-CoV-2 health related behaviors.
  Interventions: Behavioral: Phase II Promotores de Salud
- Active Comparator, Residential density-located venue placement strategy (Experimental): This is the Phase I intervention (Clinical Trial ID: NCT04793464). It includes the Phase I Promotores de Salud intervention, which consists of outreach to promote testing and vaccination at re-occurring testing events that have been selected for sites that have a high residential density of Latinx persons. At the testing events, it includes the on-site Promotores de Salud psychoeducation related to SARS-CoV-2 health related behaviors.
  Interventions: Behavioral: Phase I Promotores de Salud Outreach

INTERVENTIONS:
Behavioral: Phase II Promotores de Salud — Community partners (e.g., Mexican Consulate) select events for testing and use their usual outreach methods to attract participants to the site and their event. Then, at the community partner's event, the research team holds COVID-19 testing events and the Promotores de Salud health behavior intervention is delivered by bilingual research staff. The health behavior intervention includes: 1) psychoeducation to promote hand-washing, social distancing, mask wearing if unvaccinated, and continued testing to mitigate the spread of COVID-19 and psychoeducation to address vaccine hesitancy; 2) information support and service navigation to address logistical challenges associated with testing and vaccination (e.g., scheduling health care visits, transportation, language barriers); 3) motivational interviewing to explore personal, social, and behavioral barriers to testing and vaccination, and to discuss available resources.
  Other Names: Phase II Outreach + Promotores on Site
  Arms: Partner-optimized venue placement strategy
Behavioral: Phase I Promotores de Salud Outreach — Testing events re-occur every two weeks at the same location and time, based on census density on Latinx individuals for site selection. Outreach conducted by promotores occurs to increase attendance at the testing events. Outreach is culturally responsive (e.g., culturally tailored radio announcements, social media posts, community canvassing, referral by community leaders).
  Other Names: Phase I Outreach
  Arms: Active Comparator, Residential density-located venue placement strategy

SUMMARY:
The global SARS-CoV-2 pandemic that causes the severe respiratory illness COVID-19 is the worst health crisis that the United States has faced in a century. Although this highly contagious virus has infected millions of Americans already, the disease burdens are disproportionately born by historically underserved populations such as Latinx communities. In Oregon, 13% of the population that is Latinx represents approximately 25.7% of COVID-19 cases and are burdened with more than twice the cases per 100,000 individuals compared to non-Hispanic Oregonians (10,677 versus 4,616, respectively). Furthermore, only 54.9% of eligible Latinx Oregonians are vaccinated compared to the 76.2% statewide vaccination rate. An urgent need exists to reach Oregon's Latinx community to prevent SARS-CoV-2 transmission and increase vaccine acceptance.

The overall goal of this study is to implement a Promotores de Salud behavioral health intervention to increase the reach, access, uptake, and impact of testing and vaccination in Latinx communities in Oregon. This project will fully integrate with the National institutes of Health (NIH) Rapid Acceleration of Diagnostics (RADx) consortium and its Coordination and Data Collection Center (CDCC). The study team will add testing venues based on feedback from the Oregon Health Authority (OHA) and our county and community partners to test if a "partner-optimized venue placement strategy" yields more Latinx individuals tested than placement of sites based upon residential density used in the ongoing testing in Phase I of this study (Clinical Trial ID: NCT04793464). In addition, evaluation of the Promotores de Salud intervention held during testing events will test whether culturally competent education results in greater use of strategies that reduce transmission of COVID-19 at the community and individual level and increases the number of individuals who choose to be vaccinated, as a function of fidelity of the intervention. Over time, this project will help communities institutionalize optimal local testing frameworks supported by University of Oregon laboratory facilities for testing capacity, technical support for testing logistics, and collection of data on health behaviors, testing rates, and sustainability. The resulting structures and systems will be poised for future scale-up to other vulnerable communities and/or for other public health purposes.

DETAILED DESCRIPTION:
This study will test, compare, and determine if targeted placement of testing events at venues identified each month as viable by the Oregon Health Authority, Community Based Organizations, and our community partners ("partner-optimized venue placement strategy") will increase the number of Latinx individuals who get tested. All testing events will receive the Promotores de Salud intervention, which includes Spanish/English bilingual community health workers (i.e., promotores) from the local communities delivering health information to everyone attending testing events.

Promotores will deliver the Promotores de Salud intervention and promote strategies that are effective in mitigating the spread of COVID-19. They will also emphasize the continued importance of preventive strategies given the increasing availability of vaccines and addressing vaccine hesitancy. This health information will be shared at testing events via brief verbal interactions and printed materials (i.e., brochures and infographics). The intervention will also specifically address logistical challenges associated with vaccination uptake (e.g., lack of transportation, language barriers, and difficulty locating vaccination opportunities), which are additional factors driving vaccine hesitancy among Latinx communities. The Promotores de Salud intervention was designed to build relationships with Latinx community members and facilitate trust.

To assess the proportion of Latinx community members tested at each site, the investigators will use de-identified health information from a patient registry provided to the study by the University of Oregon's (UO) COVID-19 clinical genomics laboratory, who are processing the tests. The investigators anticipate engaging a greater proportion of Latinx community members, relative to overall county demographics, at the testing events. The investigators also expect to enroll more proportionally more Latinx individuals as these events, relative to Phase I events. The overall study population is expected to be 75% Hispanic and 25% non-Hispanic, with 87% of individuals identifying as White in both ethnic groups and the remaining 13% identifying as African American, Asian, Pacific Islander, American Indian/Alaska Native, or more than one race. The investigators anticipate testing approximately 100 people per month, across 11 months and 24 events, for a total of 1,100 individuals tested. To assess health behaviors, a subset of adult participants at each testing event will be invited to participate in a research survey, administered at testing (baseline) and again 30 days later (T2). Of the 1,100 individuals tested, the team anticipates that 50% will choose to participate in the research survey for a total of 550 individual participants. Survey data from baseline to T2 will be used to examine the effectiveness of the promotores intervention, as a function of intervention fidelity.

Quality Assurance, Data Checks, Source Data Verification, Data Dictionary, and Standard Operating Procedures: Data and biospecimens will be collected in-person at testing sites, requiring direct interaction with participants. In order to report SARS-CoV-2 infection results back to each participant, name, date of birth, and contact information are collected. To fulfill reporting requirements to the Oregon Health Authority, county of residence and zip code are also collected for each person tested. Data used to evaluate the efficacy of intervention will involve aggregate variables derived from data collected as part of the diagnostic testing procedure and will be aggregated at the level of the testing site (e.g., tests performed, race and ethnicity percentages, etc.).

For the collection of SARS-CoV-2 samples, testing facilitators will guide participants in the self-collection process. For anterior nares, participants are instructed to place the nasal swab about 1cm into their nostril and rotate it, making contact with the nasal membrane for 10 seconds, then repeating the process with the same swab in the other nostril. Testing site staff can assist participants who have low dexterity or physical impairments in sample collection. In case of an injury during sample collection, the partnering community organization staff will direct the participant to the appropriate medical resources. Samples will be placed into sterile barcoded vials (1 ml Matrix, barcoded screw-cap tubes) that each contain 500 microliters (μl) of DNA/RNA Shield. Each Matrix tube will then be closed tightly and will be placed in a standard plastic laboratory microcentrifuge tube rack with eight rows and twelve columns (8-by-12 rack with 96 positions). This rack will then be externally decontaminated by brief submersion in accelerated hydrogen peroxide (H202). Each 96-position microcentrifuge tube rack will then be labeled and placed in a sterile temporary container with an icepack. At the end of the day all racks will be transported to the COVID-19 clinical genomics Laboratory at UO, ensuring that they will arrive no longer than 48 hours after collection.

Each 96 well collection plate will next proceed to molecular processing using the standard, FDA approved Thermo Fisher TaqPath or Diacarta Quantivirus analysis protocols, which are similar nucleic acid amplification tests (NAAT). All steps of this approved protocol will be followed exactly, including the appropriate reagents, volumes, inclusion of appropriate positive and negative controls and the software analysis system and parameters. Hamilton liquid handling robots (Hamilton, Microlab VANTAGE 2.0) are used to aliquot from 96 tube matrix racks and for subsequent qPCR amplification. All laboratory assays and reporting will be automated through the use of barcodes, robotics, 96 and 384 well qPCR machines, and the use of a fully HIPAA and CAP3 compliant Laboratory Information Management System (LIMS) built by L7 informatics (https://l7informatics.com/), which organizes and relays information from lab instruments to secure databases. The results for each sample, and associated metadata, are then associated with each assigned barcode and can then be disseminated, as appropriate, to the Oregon Health Authority, the appropriate county health department, and the individual. Test results will be available within 48 hours and no later than 4 days to the individual and/or the health authority. After testing occurs, researchers will have access to aggregate, community-level (e.g., counts and prevalence rates), de-identified data prepared by the data managers in collaboration with the UO's CLIA clinical genomics laboratory. The data will include three protected health identifiers: site zip code, participant zip code, and testing date. It will also include demographic data this is not protected health information such as age range, race, and ethnicity. These data will be used to assess outreach activities aimed at increasing participation of Latinx community members in SARS-COV-2 testing. The primary outcome for this aspect of the study is site-level testing rates of Latinx individuals.

Sample Size Assessment, Plan for Missing Data, Statistical Analysis Plan: To test the hypothesis that partner-optimized venue placement (Phase II) yields more Latinx individuals tested than placement of sites based upon residential density (Phase I), analyses will employ comparative effectiveness research approaches (CER) using a clustered quasi-experimental comparison of our implementation outreach. These analyses comprise two study arms to compare the number of Latinx tested between top-performing Phase I sites (census geo-located venue placement) contrasted with Phase II (partner-optimized venue placement). The primary outcome for partner-optimized venue placement will be the number of Latinx tested specified as a generalized linear multilevel count of test samples collected, nesting events over time within site locations. To address internal validity threats to the quasi-experimental design, study investigators will employ propensity score matching procedures for all pooled data analyses comparing the two conditions. Primary analyses are powered to detect medium effects.

To test the hypothesis that accurate and culturally tailored information delivered by promotores at testing events will result in individual level outcomes, study investigators will evaluate whether implementation fidelity of the Promotores de Salud health intervention will improve testing, reduce vaccination hesitancy, and increase vaccine acceptance and improve health literacy. Social determinants of testing and vaccination analyses will focus on the contextual determinants of pre-post change in the likelihood of vaccination, repeated testing for those unvaccinated, and reduced vaccine hesitancy. Analyses will focus on within-intervention group pre-post change specified as linear mixed models for vaccine hesitancy and generalized linear mixed models for testing counts and vaccine acceptance. These analyses are powered to detect small to moderate effects.

Two primary sources of missing data are expected, item non-response and attrition over time. For dropout, investigators will conduct standard attrition analyses to compare baseline characteristics between attriters and completers. They will consider propensity score matching procedures and complier average causal effects models to address substantial differences. For item non-response and scale score development, investigators will require 70% of scale items be present for scoring. They will test whether scale level data are missing completely at random (MCAR) within waves and then across waves. If data are not MCAR, under assumptions of missing at random (MAR, i.e., data are not dependent on missing values of the intervention response variable), investigators will employ one of two recommended approaches for SEM, full information maximum likelihood (FIML) or multiple imputation (MI). Although these approaches can be problematic when data are non-ignorable missing, they are still recommended for handling missingness, particularly with covariates associated with attrition. Both methods provide more efficient standard errors than listwise or pairwise deletion, or mean substitution. Should missing data or attrition be associated with covariates, investigators will include appropriate covariates in hypothesis testing.

Finally, data will be collected in accordance with Tier 1 "common data elements" from the national Duke Coordination and Data Collection Center (CDCC). The CDCC directly assists each individual RADx-UP project to optimize engagement, outreach, testing strategies, and to facilitate co-learning opportunities between and among RADx-UP projects. Key outcome data and the testing procedures for obtaining the sample, analysis platform, analysis procedures, and test resulting will be collected and represented in a consistent manner for harmonization across the consortium, integrated with test reporting requirements under the Coronavirus Aid, Relief, and Economic Security Act (CARES Act).

ELIGIBILITY:
Inclusion Criteria:

* Proportion Tested: Age 3 or older
* Proportion Tested: Received testing at study testing site
* Individual Survey: 15 or older

Exclusion Criteria:

• Individual Survey: Unable to understand Spanish or English or another language translated by a qualified translator at a 5th grade level

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1463 (Actual)
Dates: Start 2021-09-15 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leslie D Leve, PhD, Principal Investigator — University of Oregon
Locations (1):
- University of Oregon, Eugene, Oregon, United States

IPD SHARING:
Plan to Share IPD: Yes
The investigators will share IPD with the RADx-Up CDCC. All Tier 1 data elements required by the CDCC will be shared, unless we receive an official exception for some items from the CDCC and NIH.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: IPD will be shared in accordance with timeframes set by the RADX-UP CDCC
Access Criteria: The RADX-UP CDCC will make these determinations
URL: http://radx-up.org/about/

REFERENCES:
- [Derived] Leve LD, DeGarmo DS, Searcy J, Budd EL, Ramirez Garcia JI, Mauricio AM, Cresko WA. Attendance of Underserved Populations at Field-Based Health Services Events: Application of Quasi-Experimental Methods that Accommodate the COVID-19 Pandemic. Prev Sci. 2025 Jan 20. doi: 10.1007/s11121-025-01769-z. Online ahead of print. PMID 39828881
- [Derived] Ramirez Garcia JI, Oro V, Budd EL, Mauricio AM, Cioffi CC, Anda S, McWhirter EH, DeGarmo DS, Leve LD. A Translational Case Study of a Multisite COVID-19 Public Health Intervention Across Sequenced Research Trials: Embedding Implementation in a Community Engagement Phased Framework. Am J Public Health. 2024 May;114(S5):S396-S401. doi: 10.2105/AJPH.2024.307669. PMID 38776498

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1463 participants enrolled in this Clinical Trial. The active comparator group was all participants enrolled in the Phase I study (Clinical Trial ID: NCT04793464).
Groups:
- Active Comparator, Residential Density-located Venue Placement Strategy: This is the Phase I study (Clinical Trial ID: NCT04793464) and is comprised of the "Promotores", "Control", and "Unknown Treatment Status" Arms/Groups from the Phase I study. For all Phase I study activities, testing events re-occurred every two weeks at the same location and time, based on census density on Latinx individuals for site selection.
  Promotores de Salud intervention arm consists of outreach to promote testing and vaccination at re-occurring testing events that have been selected for sites that have a high residential density of Latinx persons. At the testing events, it includes the on-site Promotores de Salud psychoeducation related to SARS-CoV-2 health related behaviors. Outreach conducted by promotores occurs to increase attendance at the testing events. Outreach is culturally responsive (e.g., culturally tailored radio announcements, social media posts, community canvassing, referral by community leaders).
  Control treatment status sites consisted of sites with "business as usual" outreach methods. No additional outreach activities were completed and promotores were not on site to deliver the Promotores de Salud intervention.
  Unknown treatment status participants had data collected at an intervention or control site, but their exposure status is unknown.
Period: Overall Study
Arm/Group | Partner-optimized Venue Placement Strategy | Active Comparator, Residential Density-located Venue Placement Strategy
Started | 1463 | 1623
Completed | 887 | 934
Not Completed | 576 | 689
Not completed — Lost to Follow-up | 549 | 631
Not completed — Withdrawal by Subject | 27 | 58

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Partner-optimized Venue Placement Strategy | Active Comparator, Residential Density-located Venue Placement Strategy | Total
Number analyzed (Participants) | 1463 | 1623 | 3086
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 40 [30 to 50] | 40 [28 to 51] | 40 [29 to 50]
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 927 | 943 | 1870
  Male | 450 | 633 | 1083
  Unknown | 86 | 47 | 133
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1177 | 1107 | 2284
  Not Hispanic or Latino | 193 | 459 | 652
  Unknown or Not Reported | 93 | 57 | 150
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 178 | 186 | 364
  Asian | 6 | 29 | 35
  Native Hawaiian or Other Pacific Islander | 7 | 10 | 17
  Black or African American | 19 | 16 | 35
  White | 185 | 423 | 608
  More than one race | 40 | 59 | 99
  Unknown or Not Reported | 1028 | 900 | 1928
Region of Enrollment [Number; unit: participants]
  United States | 1463 | 1623 | 3086
Testing Barriers and Hesitancy [Mean (Standard Deviation); unit: units on a scale] — This measure is built around the following question: "Did you have any of the following concerns or face any of the following challenges when deciding to get tested today? Select all that apply." Participants are asked to indicate 'yes', 'somewhat', or 'no' in response to a list of 13 options. Mean ranges from 0-2 with higher scores indicating a higher number of barriers faced. This measure is adapted from the paper Development and psychometric testing of a barriers to HIV testing scale among individuals with HIV infection in Sweden; The Barriers to HIV testing scale-Karolinska version. Population: Number analyzed is the number of participants with valid baseline data.
  units on a scale
    number analyzed (Participants) | 1021 | 339 | 1360
    (all) | 0.34 (0.45) | 0.39 (0.43) | 0.35 (0.45)
Vaccination Attitudes Examination (VAX) Scale [Mean (Standard Deviation); unit: units on a scale] — Participants are asked to rate their agreement (6-point Likert scale: strongly agree to strongly disagree) on 15 qualitative statements about vaccinations. For example, "I feel safe after being vaccinated" and "Vaccination programs are a big con." Means range from 1-6 with higher scores associating with higher vaccination acceptance. Population: Number analyzed is the number of participants with valid baseline data.
  units on a scale
    number analyzed (Participants) | 1116 | 353 | 1469
    (all) | 3.45 (1.01) | 3.50 (0.94) | 3.46 (0.99)
COVID-19 Prevention Health Behaviors [Mean (Standard Deviation); unit: units on a scale] — From the PhenX toolkit, Protocol - COVID-19 Knowledge, Attitudes, and Avoidant Behaviors, participants are asked to indicate "Which of the following have you done in the last seven days to keep yourself safe from coronavirus? Only consider actions that you took or decisions that you made personally." There are a total of 3 possible items participants rate as a binary, Yes/No, response. The count of 'yes' responses was recorded. The scale will range from 0-3. A higher score indicates more preventative behaviors. Population: Number analyzed is the number of participants with valid baseline data.
  units on a scale | 2.3 (0.9) | 2.4 (0.8) | 2.4 (0.8)
COVID-19 Knowledge and Attitudes 1 [Mean (Standard Deviation); unit: units on a scale] — Participants were asked: "In your opinion, how effective are the following actions for keeping you safe from COVID-19?" A list of 3 prevention strategies are listed. Participants indicate their response on a scale Very Effective (5) to Not Effective at AlI (1). Scale range is 1-5. A mean value is computed. Higher scores indicate a better outcome. Population: Number analyzed is the number of participants with valid baseline data.
  units on a scale
    number analyzed (Participants) | 1360 | 1554 | 2914
    (all) | 4.2 (0.9) | 4.2 (0.8) | 4.2 (0.9)
COVID-19 Knowledge and Attitudes 2 [Mean (Standard Deviation); unit: units on a scale] — Participants were asked: "How safe or unsafe are the following actions for avoiding exposure to coronavirus?" A list of 3 activities are listed and responses are on scale of 1 (Extremely Unsafe) to 4 (Extremely Safe). Mean scores were calculated. Scores range between 1-4. Higher score means a worse outcome. Population: Number analyzed is the number of participants with valid baseline data.
  units on a scale
    number analyzed (Participants) | 1266 | 1473 | 2739
    (all) | 2.2 (0.8) | 2.0 (0.7) | 2.1 (0.7)

OUTCOME MEASURES:

1. Primary Outcome: Testing Barriers and Hesitancy
Description: This measure is built around the following question: "Did you have any of the following concerns or face any of the following challenges when deciding to get tested today? Select all that apply." Participants are asked to indicate 'yes', 'somewhat', or 'no' in response to a list of 13 options. Scale ranges from 0-2 with higher scores indicating a higher number of barriers faced. This measure is adapted from the paper Development and psychometric testing of a barriers to HIV testing scale among individuals with HIV infection in Sweden; The Barriers to HIV testing scale-Karolinska version (Wiklander et al., 2015).
Time Frame: Change from baseline to 30 days
Population: Number analyzed is the number of participants with valid baseline and follow-up data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Partner-optimized Venue Placement Strategy | Active Comparator, Residential Density-located Venue Placement Strategy
Number analyzed (Participants) | 549 | 169
score on a scale | 0.29 (0.38) | 0.24 (0.34)
Statistical Analysis 1: Comparison: Partner-optimized Venue Placement Strategy vs Active Comparator, Residential Density-located Venue Placement Strategy; Test type: Superiority; p = 0.09, ANCOVA; Mean Difference (Final Values) = 0.048, 95% CI 2-sided [-0.008 to 0.104]

2. Primary Outcome: Vaccination Attitudes Examination (VAX) Scale
Description: Participants are asked to rate their agreement (6-point Likert scale: strongly agree to strongly disagree) on 15 qualitative statements about vaccinations. For example, "I feel safe after being vaccinated" and "Vaccination programs are a big con." Means range from 1-6 with higher scores associating with higher vaccination acceptance. This measure is adapted from the VAX Scale (Martin et al., 2017).
Time Frame: Change from baseline to 30 days
Population: Number analyzed is the number of participants with valid baseline and follow-up data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Partner-optimized Venue Placement Strategy | Active Comparator, Residential Density-located Venue Placement Strategy
Number analyzed (Participants) | 607 | 175
score on a scale | 3.58 (0.82) | 3.44 (0.72)
Statistical Analysis 1: Comparison: Partner-optimized Venue Placement Strategy vs Active Comparator, Residential Density-located Venue Placement Strategy; Test type: Superiority; p = 0.02, ANCOVA; Mean Difference (Final Values) = 0.15, 95% CI 2-sided [0.02 to 0.29]

3. Primary Outcome: COVID-19 Prevention Health Behaviors
Description: From the PhenX toolkit, Protocol - COVID-19 Knowledge, Attitudes, and Avoidant Behaviors, participants are asked to indicate "Which of the following have you done in the last seven days to keep yourself safe from coronavirus? Only consider actions that you took or decisions that you made personally." There are a total of 3 possible items participants rate as a binary, Yes/No, response. The count of 'yes' responses are recorded. The scale will range from 0-3. A higher score indicates more preventative behaviors.
Time Frame: Change from baseline to 30 days
Population: Number analyzed is the number of participants with valid baseline and follow-up data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Partner-optimized Venue Placement Strategy | Active Comparator, Residential Density-located Venue Placement Strategy
Number analyzed (Participants) | 887 | 934
score on a scale | 2.3 (0.8) | 2.4 (0.7)
Statistical Analysis 1: Comparison: Partner-optimized Venue Placement Strategy vs Active Comparator, Residential Density-located Venue Placement Strategy; Test type: Superiority; p = 0.03, ANCOVA; Ratio of Means = -0.076, 95% CI 2-sided [-0.145 to -0.007]

4. Primary Outcome: COVID-19 Knowledge and Attitudes 1
Description: Participants were asked: "In your opinion, how effective are the following actions for keeping you safe from COVID-19?" A list of 3 prevention strategies are listed. Participants indicate their response on a scale Very Effective (5) to Not Effective at AlI (1). Scale range is 1-5. A mean value is computed. Higher scores indicate a better outcome.
Time Frame: Change from baseline to 30 days
Population: Number analyzed is the number of participants with valid baseline and follow-up data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Partner-optimized Venue Placement Strategy | Active Comparator, Residential Density-located Venue Placement Strategy
Number analyzed (Participants) | 831 | 901
score on a scale | 4.2 (0.8) | 4.2 (0.7)
Statistical Analysis 1: Comparison: Partner-optimized Venue Placement Strategy vs Active Comparator, Residential Density-located Venue Placement Strategy; Test type: Superiority; p = 0.38, ANCOVA; Mean Difference (Final Values) = 0.03, 95% CI 2-sided [-0.04 to 0.09]

5. Primary Outcome: COVID-19 Knowledge and Attitudes 2
Description: Participants were asked: "How safe or unsafe are the following actions for avoiding exposure to coronavirus?" A list of 3 activities are listed and responses are on scale of 1 (Extremely Unsafe) to 4 (Extremely Safe). Mean scores were calculated. Scores range between 1-4. Higher score means a worse outcome.
Time Frame: Change from baseline to 30 days
Population: Number analyzed is the number of participants with valid baseline and follow-up data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Partner-optimized Venue Placement Strategy | Active Comparator, Residential Density-located Venue Placement Strategy
Number analyzed (Participants) | 759 | 837
score on a scale | 2.2 (0.7) | 2.0 (0.6)
Statistical Analysis 1: Comparison: Partner-optimized Venue Placement Strategy vs Active Comparator, Residential Density-located Venue Placement Strategy; Test type: Superiority; p = 0.002, ANCOVA; Mean Difference (Final Values) = 0.096, 95% CI 2-sided [0.04 to 0.16]

ADVERSE EVENTS:
Time Frame: Adverse events were monitored/assessed through study completion, approximately 6 months.
Arm/Group | Partner-optimized Venue Placement Strategy | Active Comparator, Residential Density-located Venue Placement Strategy
All-Cause Mortality (participants affected / at risk) | 0/1463 | 0/1623
Serious Adverse Events (participants affected / at risk) | 0/1463 | 0/1623
Other Adverse Events (participants affected / at risk) | 0/1463 | 0/1623

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2021-11-15): https://cdn.clinicaltrials.gov/large-docs/35/NCT05082935/Prot_001.pdf
  • Statistical Analysis Plan (2021-05-27): https://cdn.clinicaltrials.gov/large-docs/35/NCT05082935/SAP_002.pdf
  • Informed Consent Form (2021-07-21): https://cdn.clinicaltrials.gov/large-docs/35/NCT05082935/ICF_000.pdf